CLINICAL TRIAL: NCT07030088
Title: Clinical and Patient-Based Evaluation of a Novel Dual-Headed Toothbrush Design: Split-Mouth Clinical Trial
Brief Title: Evaluation of a Novel Dual-Headed Toothbrush Design for Periodontal Health: Split-Mouth Randomized Blind Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dar Al Uloom University (Other)
Responsible Party: Principal Investigator, Sally Abd-ElMeniem ElHaddad, Assist. Prof. Periodontology and Oral Medicine, Dar Al Uloom University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 34-01-2025
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-06

CONDITIONS: Dental Plaque Accumulation; Oral Hygiene Education Methods; Toothbrushing
Keywords: Dual-headed toothbrush; Single-headed toothbrush; Toothbrushing technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-Headed Toothbrush (Experimental): Participants used a dual-headed manual toothbrush to clean one side of their mouth (maxillary and mandibular quadrants). Brushing was performed using the Bass technique, twice daily. This arm assesses the effectiveness, comfort, and time-efficiency of the novel dual-headed toothbrush design.
  Interventions: Device: Dual-Headed Manual Toothbrush
- Single-Headed Toothbrush (Active Comparator): Participants used a conventional single-headed manual toothbrush to clean the other side of their mouth using the same brushing technique (Bass method), frequency (twice daily). This arm serves as the standard control for comparison in evaluating plaque removal and patient-reported comfort.
  Interventions: Device: Conventional Single-Headed Manual Toothbrush

INTERVENTIONS:
Device: Dual-Headed Manual Toothbrush — A novel toothbrush with a dual-headed design intended to clean both upper and lower buccal/ or upper and lower lingual/ palatal surfaces simultaneously. Participants were instructed to use this toothbrush on one side of the mouth only, twice daily using the Bass brushing technique. This intervention is evaluated for plaque removal efficacy, gingival health, brushing time, and patient comfort
  Arms: Dual-Headed Toothbrush
Device: Conventional Single-Headed Manual Toothbrush — A standard single-headed manual toothbrush used as the active control. Participants used this toothbrush on the other side of the mouth, with the same brushing technique (Bass method), frequency (twice daily). It serves as the comparator for assessing the performance of the dual-headed design.
  Arms: Single-Headed Toothbrush

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and patient satisfaction of a novel dual-headed toothbrush design compared to a conventional single-headed toothbrush in adult dental professionals aged 22-45 years with healthy gingival conditions. The main questions it aims to answer are:

Does the dual-headed toothbrush improve plaque removal efficiency compared to a single-headed toothbrush? Does the dual-headed toothbrush enhance brushing comfort, reduce brushing time, and improve user satisfaction? Researchers will compare the side of the mouth (cleaned with a dual-headed toothbrush) with the other side (cleaned with a single-headed toothbrush) in a randomized split-mouth design to see if the novel design leads to superior plaque control and better user experience.

Participants will:

Receive both toothbrush types (medium bristle) and identical toothpaste Be trained in the Bass brushing technique Use each toothbrush, twice daily, with the assigned toothbrush applied to its designated side of the mouth

Complete post-trial questionnaires on comfort, ease of use, and brushing time

DETAILED DESCRIPTION:
This clinical trial explores the comparative effectiveness and user experience of a novel dual-headed toothbrush design versus a conventional single-headed toothbrush using a randomized split-mouth methodology among adult dental professionals. Dental professionals were selected as participants due to their consistent oral hygiene habits and ability to comply with standardized brushing protocols.

The study investigates whether the dual-headed design can offer improved plaque removal efficiency, reduced brushing time, and greater comfort during use-factors that are increasingly relevant to both clinical performance and patient compliance in oral hygiene tools. Participants were trained to use both toothbrushes following the Bass technique and instructed to brush twice daily, with the left and right sides of the mouth assigned to different brushes.

The trial design allows for within-subject comparison, minimizing confounding variables such as brushing technique, motivation, and dietary habits. In addition to clinical measurements, participants' subjective experiences were captured through structured questionnaires focusing on comfort, ease of maneuverability, and time spent brushing.

This investigation aims to provide evidence to guide the development of more ergonomic and time-efficient toothbrush designs that improve plaque control without compromising user comfort. Findings from this study may influence the recommendation of dental hygiene tools, particularly for individuals seeking more efficient oral hygiene practices or patients with limited dexterity or who rely on caregivers.

ELIGIBILITY:
Inclusion Criteria:

* • Dentists with a minimum of 26 natural teeth, good general health, and the ability to perform routine oral hygiene independently.

  * No systemic diseases affecting oral hygiene.
  * Record of mild-to-moderate plaque accumulation; PI score ≥ 1
  * Rt handed dentists

Exclusion Criteria:

* • Participants with active periodontal disease, orthodontic appliances, or having recent oral surgery

  * Those currently enrolled in any other dental trial
  * Smokers.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Plaque Index (PI) | After 2, and 4 weeks of brushing
  Difference in plaque scores between baseline and end of study on the left and right sides of the mouth, using the Silness and Löe Plaque Index.
  Scale:
  0 = No plaque, 1 = A film of plaque, 2 = Moderate plaque, 3 = Abundant plaque Interpretation: Lower scores indicate better oral hygiene and effectiveness of the toothbrush.
Gingival Index (GI) | after 2 and 4 weeks
  Löe & Silness for GI Gingival index 0: Healthy gums. Gingival index 1: Mild discolouration and oedematous gingiva. No bleeding on probing.
  Gingival index 2: Red, oedematous and shiny gingiva. There is bleeding on probing.
  Gingival index 3: Red, oedematous and ulcerated gingiva. There is spontaneous bleeding.
  Interpretation: Lower scores indicate better oral hygiene and effectiveness of the toothbrush.
mSBI (modified sulcular bleeding index) | after 2, and 4 weeks
  mSBI (modified sulcular bleeding index): 0: no bleeding when a periodontal probe is passed along the gingival margin
  1. isolated bleeding spots visible
  2. Blood forms a confluent red line on margin
  3. Heavy or profuse bleeding
  Interpretation: Lower scores indicate better oral hygiene and effectiveness of the toothbrush.

SECONDARY OUTCOMES:
Brushing Time Per Side | Self-reported after 4 weeks
  Measure: Average time (in seconds) participants took to brush each side (left and right) during the trial.
  Interpretation: Shorter brushing time with equal or better plaque control is considered a favorable outcome.
Patient satisfaction and comfort | after 4 weeks
  Patient satisfaction and comfort (evaluated using a Likert scale questionnaire):
  5- point Likert scale: How easy or difficult is it to use the novel toothbrush?
  Very difficult, Somewhat difficult , Neither difficult nor easy , Somewhat easy , Very easy

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Dar AlUloom University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified individual participant data (IPD) will be made available for research purposes:
  Demographic data: Age, gender, and handedness (for brushing consistency)
  Plaque Index scores: Baseline and post-intervention scores for both left and right sides
  Brushing time data: Self-reported average brushing time per side
  Toothbrush preference: Participant-reported final preference (dual-headed vs. single-headed)
Supporting Information: Study Protocol, ICF, CSR